CLINICAL TRIAL: NCT02603081
Title: Phase 1b Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of SPI-1005 in Meniere's Disease
Brief Title: Study to Evaluate SPI-1005 in Adults With Meniere's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sound Pharmaceuticals, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPI-1005-151
Record Dates: First submitted 2015-11-02; First posted 2015-11-11 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Meniere's Disease
Keywords: Meniere's; hearing loss; vertigo; tinnitus; ebselen
MeSH Terms: conditions — Meniere Disease; Hearing Loss; Vertigo; Tinnitus | interventions — ebselen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): 0 mg SPI-1005 bid po x 21d
  Interventions: Drug: SPI-1005
- Low dose (Active Comparator): 200 mg SPI-1005 bid po x 21d
  Interventions: Drug: SPI-1005
- Mid dose (Active Comparator): 400 mg SPI-1005 bid po x 21d
  Interventions: Drug: SPI-1005
- High dose (Active Comparator): 600 mg SPI-1005 bid po x 21d
  Interventions: Drug: SPI-1005

INTERVENTIONS:
Drug: SPI-1005 — Ebselen is a small molecule mimic and inducer of glutathione peroxidase (GPx). GPx reduces reactive oxygen species by the binding of free radicals to its selenium moiety. Ebselen has strong anti-inflammatory characteristics.
  Other Names: ebselen

SUMMARY:
This study will evaluate the safety and efficacy of three dose levels of SPI-1005 compared to placebo on vertigo, tinnitus and sensorineural hearing loss in 40 adults with Meniere's disease.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled safety, pharmacokinetic, pharmacodynamic study of oral SPI-1005 in adults with Meniere's disease. All subjects will undergo baseline audiometric testing and have their severity of sensorineural hearing loss, tinnitus and vertigo determined before the start of a 21-day course of treatment with SPI-1005 or placebo. During treatment with SPI-1005, and 7 days and 28 days following the cessation of SPI-1005, subjects will have their hearing loss, tinnitus and vertigo assessed. Additional testing including electrocochleography will be performed at baseline, at the end of SPI-1005 treatment, and 28 days after the SPI-1005 treatment has stopped. Six outpatient visits will be performed over a 7-week period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable or definite Meniere's Disease by AAO-HNS 1995 criteria within 12 months of study enrollment;
* Voluntarily consent to participate in the study;
* Females of childbearing potential should be using and committed to continue using one of the following acceptable birth control methods:

  * Sexual abstinence (inactivity) for 14 days prior to screening through study completion; or
  * IUD in place for at least 3 months prior to study through study completion; or
  * Barrier method (condom or diaphragm) with spermicide for at least 14 days prior to screening through study completion; or
  * Stable hormonal contraceptive for at least 3 months prior to study through study completion; or
  * Surgical sterilization (vasectomy) of partner at least 6 months prior to study.
* Females of non-childbearing potential should be surgically sterile (bilateral tubal ligation with surgery at least 6 months prior to study, hysterectomy, or bilateral oophorectomy at least 2 months prior to study) or be at least 3 years since last menses.

Exclusion Criteria:

* Current use or within 90 days prior to study of ototoxic medications such as aminoglycoside antibiotics (gentamicin, tobramycin, amikacin, streptomycin); platinum-containing chemotherapies (cisplatin, carboplatin, oxaliplatin); or loop diuretic (furosemide);
* History of idiopathic sensorineural hearing loss, otosclerosis, or vestibular schwannoma;
* History of middle ear or inner ear surgery;
* Current conductive hearing loss or middle ear effusion;
* Significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, or psychiatric disease;
* History of hypersensitivity or idiosyncratic reaction to compounds related to ebselen;
* Current use or within 30 days prior to study of drugs or substances known to be strong inhibitors or inducers of cytochrome P450 enzymes;
* Participation in another investigational drug or device study within 90 days prior to study enrollment;
* Female patients who are pregnant or breastfeeding.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-12; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of SPI-1005 using histories, physical exams, and clinical measures. | 7 weeks
  Incidence of of Treatment-Emergent Adverse Events

SECONDARY OUTCOMES:
Plasma Ebselen levels of SPI-1005 before, during, and after 21 days of dosing | 7 weeks
  Evaluation of potential accumulation of study drug
Plasma Selenium levels before, during, and after 21 days of dosing | 7 weeks
  Evaluation of potential changes in plasma selenium levels
Impact on Sensorineural Hearing Loss | 7 weeks
  Pure Tone Audiometry
Impact on Speech Discrimination | 7 weeks
  Words in Noise Test
Impact on Tinnitus | 7 weeks
  Questionnaire
Impact on Vertigo | 7 weeks
  Questionnaire
Pharmacodynamic response | 7 weeks
  Electrocochleography

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Kil, MD, Study Chair — Sound Pharmaceuticals
Locations (5):
- United States (5):
  - House Clinic, Los Angeles, California
  - New York Otology, New York, New York
  - MUSC, Charleston, South Carolina
  - Sound Pharmaceuticals, Inc., Seattle, Washington
  - Northwest Ear, Seattle, Washington

REFERENCES:
- [Background] Kil J, Pierce C, Tran H, Gu R, Lynch ED. Ebselen treatment reduces noise induced hearing loss via the mimicry and induction of glutathione peroxidase. Hear Res. 2007 Apr;226(1-2):44-51. doi: 10.1016/j.heares.2006.08.006. Epub 2006 Oct 6. PMID 17030476
- [Background] Lynch E, Kil J. Development of ebselen, a glutathione peroxidase mimic, for the prevention and treatment of noise-induced hearing loss. Semin Hear 2009; 30(1):47-55.
- [Background] Kil J, Harruff EE, Longenecker RJ. Development of ebselen for the treatment of sensorineural hearing loss and tinnitus. Hear Res. 2022 Jan;413:108209. doi: 10.1016/j.heares.2021.108209. Epub 2021 Feb 19. PMID 33678494
- [Derived] Garland M, Hryckowian AJ, Tholen M, Bender KO, Van Treuren WW, Loscher S, Sonnenburg JL, Bogyo M. The Clinical Drug Ebselen Attenuates Inflammation and Promotes Microbiome Recovery in Mice after Antibiotic Treatment for CDI. Cell Rep Med. 2020 Apr 21;1(1):100005. doi: 10.1016/j.xcrm.2020.100005. PMID 32483557